CLINICAL TRIAL: NCT02134782
Title: A Randomized Controlled Trial of Individualized Yoga to Reduce Fatigue in Hospitalized Children Receiving Intensive Chemotherapy
Brief Title: Yoga Fatigue Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed early for poor accrual when 125/210 planned participants had been enrolled and randomized to yoga (n=62) or iPad (n=63).
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Pediatric Oncologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Yoga RCT
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia in Relapse; Burkitt's Lymphoma Stage III; Burkitt's Lymphoma Stage IV; Type 3 Diffuse Large B-Cell Lymphoma
Keywords: Randomized Controlled Trial, yoga, children, chemotherapy, haematopoietic stem cell transplantation, fatigue, quality of life
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized Yoga Intervention Group (Experimental): Yoga will be administered individually by a trained yoga instructor, and offered daily for 21 days (5 days per week or 15 days in total). There will be a common structure for all sessions that will include relaxation and breathing exercises. Additional poses focused on strength, flexibility, and balance will be incorporated at low, moderate or high intensity levels based upon the wishes and abilities of the child and parent and the judgment of the yoga instructor. The target intensity will be documented and may change with each yoga session. Each yoga session will vary in duration between 15 and 45 minutes. Modifications will be made to accommodate devices such as central venous lines, particularly if accessed. For children who are in isolation, the research team will follow hospital policies and procedures.
  Interventions: Behavioral: Individualized Yoga Intervention Group
- iPad Activity Control Group (Active Comparator): For those randomized to the control group, visits by the same yoga instructors will occur at the same schedule as the yoga intervention. Contact will be offered daily (5 days per week) for 21 days. The yoga instructor will offer games, music, movies or books on a study-supplied iPad. The instructor will offer to interact with the child (for example, read to, or play games with the child) for a maximum of 45 minutes (the maximum length of yoga sessions). This approach will allow us to control for contact frequency and the individual providing contact, and consequently, to better measure the independent effect of yoga. These children will not receive yoga during the 3 week iPad activity period; instructors will receive specific training to ensure that no yoga occurs during this time frame. Use of child or hospital supplied iPad activities will be permitted instead of the study-supplied iPad activities.
  Interventions: Other: iPad Activity Control Group

INTERVENTIONS:
Behavioral: Individualized Yoga Intervention Group — These children will not receive a study-supplied iPad. Use of child or hospital supplied iPad games, music, movies or books will be permitted without any modification, encouragement or discouragement of these activities. There will be no restrictions on concomitant medications. Standardized sleep hygiene recommendations will be provided.
  Arms: Individualized Yoga Intervention Group
Other: iPad Activity Control Group — These children will not receive yoga during the 3 week iPad activity period; instructors will receive specific training to ensure that no yoga occurs during this time frame. Use of child or hospital supplied iPad activities will be permitted instead of the study-supplied iPad activities. There will be no restrictions on concomitant medications. Standardized sleep hygiene recommendations will be provided.
  Arms: iPad Activity Control Group

SUMMARY:
Fatigue is a major problem in children, adolescents and adults receiving intensive chemotherapy for cancer and in patients undergoing hematopoietic stem cell transplantation (HSCT). Guidelines from the National Comprehensive Cancer Network suggest that all patients, including children as young as 5 years of age, should be routinely screened for fatigue at the initial visit and at regular intervals throughout and following anti-cancer treatment. These guidelines also suggest that fatigue should be managed according to clinical practice guidelines. However, evidence demonstrating effective interventions for fatigue in children with cancer is scarce. Exercise is an effective intervention for cancer-related fatigue in patients of all ages. However, patients receiving the most intensive treatments may be too ill to participate in a standardized exercise program. A unique and potentially effective intervention that combines exercise and relaxation is yoga. This randomized controlled trial (RCT) will determine whether a 3 week program of individualized yoga is associated with less fatigue, better quality of life (QoL) and less systemic opioid use compared to the control program of an Apple tablet (iPad) games, music, movies or books. This is a multi-center, parallel-group, randomized trial of individualized yoga for fatigue. Subjects are inpatients 8-18 years of age receiving intensive chemotherapy for cancer or undergoing HSCT who are expected to remain in hospital for 3 weeks. Participants will be randomized to the individualized yoga program or to the iPad activity control program. For those who remain hospitalized on day 21, the alternate intervention will be offered for 1 week and the preferred strategy will be determined. Yoga has the potential to significantly reduce fatigue, a prevalent and distressing symptom, in children with cancer and HSCT. The investigators have assembled the optimal team with the expertise and track record to accomplish this important trial. This trial is an incremental and critically important step in a program of research designed to improve health for children at the highest risk for poor quality of life. Results may have broad applicability to other hospitalized pediatric populations and has the potential to change in-hospital care for these patients.

DETAILED DESCRIPTION:
Background: Fatigue or tiredness is a major problem in children, adolescents and adults receiving intensive chemotherapy for cancer and in those undergoing hematopoietic stem cell transplantation (HSCT). While exercise is good for reducing fatigue, these patients are often too sick to participate in regular exercise sessions. A unique, potentially effective type of exercise is individualized yoga. Yoga is particularly good since it can be tailored to be more or less intensive depending on how the child is feeling. The investigators have previously performed a feasibility study of yoga in children admitted to the hospital receiving very intensive chemotherapy or HSCT and found that our program of yoga is doable. The investigators also found children and their parents like the program.

Preliminary Data: The investigators' team completed a feasibility study of yoga in 11 children with cancer or HSCT recipients meeting similar eligibility criteria as the proposed study. In short, these results demonstrated the feasibility of individualized yoga and suggested several design changes to enhance compliance with outcome ascertainment. The investigators found that the mean ± standard deviation for the baseline and day 21 proxy-report PedsQL MFS general fatigue scores were 46.4±26.8 and 55.6±15.5. These scores are much lower compared to fatigue scores observed in two studies of healthy children in which scores of 88.8±12.3 and 89.3±13.3 were described. This data suggest that fatigue is expected to be very severe in our patient population.

Objectives: Primary: To determine if a 3 week program of individualized yoga for hospitalized children receiving intensive chemotherapy is associated with lower general fatigue or tiredness compared to the control intervention of iPad games, music, movies or books. Secondary: To determine if a 3 week program of yoga is associated with better quality of life and less pain medication use when compared to an iPad activity control program.

Methods: This is a multi-center, randomized trial of individualized yoga for fatigue. Participants are children 8-18 years of age receiving intensive chemotherapy for cancer or undergoing HSCT who are expected to remain in hospital for 3 weeks. Participants will be randomized to individualized yoga or to the iPad activity control program. The intervention is an individualized yoga program in which intensity level may change with each session. The control program consists of visits in which games, music, movies or books on a study-supplied iPad will be offered. Yoga sessions will be offered five times a week over 3 weeks and will be led by a trained yoga teacher. In the control arm, the yoga teacher will visit once a day and will offer children games, music, movies or books on an iPad. Fatigue and quality of life will be measured by the parent at baseline, on day 10 and on day 21. For subjects who remain hospitalized on day 21, they will be offered the alternate arm for one week to promote retention.

The investigators intend to record 20% of yoga and iPad sessions using the iPad to ensure quality control and monitoring of sessions. Recorded files will be downloaded to a secure File Transfer Protocol (FTP) site. Any deviations from the protocol will result in feedback to the site within 1 week of the session and ideally, within 2 days. The research team will also routinely audit the data submitted to ensure completeness of the data submissions.

The investigators plan to enroll 210 subjects at 2 centres in Canada and 1 centre in the United States over 4 years.

Significance: Yoga has the potential to significantly reduce fatigue, a prevalent and distressing symptom, in children with cancer and HSCT. The investigators have assembled the optimal team with the expertise and track record to accomplish this important trial. This trial is an incremental and critically important step in a program of research designed to improve health for children at highest risk for poor quality of life. Results may have broad applicability to other hospitalized pediatric populations and has the potential to change in-hospital care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosed with any AML, relapsed ALL, stage 3 or 4 Burkitt's or diffuse B large cell lymphoma/leukemia OR about to receive autologous or allogeneic HSCT for any indication
* Child expected to be an inpatient for at least 3 weeks after initiation of chemotherapy or conditioning
* Child aged 8 to 18 years at enrollment. Conditioning regimen may be myeloablative or reduced intensity

Exclusion Criteria:

* Following features present to an extent that would preclude compliance with yoga, as assessed by the attending physician: a) motor disability, b) cognitive disability, c) cardiopulmonary symptoms, or d) known compression fracture resulting in disability
* Parent or patient cannot understand verbal English
* For HSCT patients, planned non-myeloablative conditioning regimen.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Change in proxy-reported general fatigue (PedsQL MFS) | Change from baseline to day 10 and day 21
  The primary outcome is parent/guardian proxy-reported general fatigue using the pediatric population validated questionnaire PedsQL Multidimensional Fatigue Scale (MFS) measured at day 21. PedsQL MFS assesses general fatigue, sleep/rest fatigue and cognitive fatigue. The investigators have chosen this fatigue measure as the primary outcome as in our experience, it is sensitive to change and it is easy to administer and complete.

SECONDARY OUTCOMES:
Change in proxy-reported other fatigue outcomes (PedsQL MFS) | Change from baseline to day 10 and day 21
  One of the secondary outcomes is the other fatigue outcomes for proxy-reported PedsQL MFS (sleep/rest fatigue and cognitive fatigue) on days 10 and 21.
Change in proxy-reported fatigue outcomes (FS-P) | Change from baseline to day 10 and day 21
  One of the secondary outcomes is the Fatigue Scale Parent (FS-P) on days 10 and 21.
Change in proxy-reported fatigue outcomes (PedsQL Acute Cancer Module) | Change from baseline to day 10 and day 21
  One of the secondary outcomes is the fatigue outcomes for proxy-reported PedsQL Acute Cancer Module (pain, nausea and anxiety) on days 10 and 21.

OTHER OUTCOMES:
Use of systemic opioids | Change from baseline to day 21
  All systemic opioid administrations between randomization and date off study will be tabulated and will be expressed as the cumulative amount in morphine equivalents/kg/day on study. Systemic opioid administration will be obtained from patient's chart review. Systemic opioid intake is o potential co-variates the could affect fatigue.
Change in self-reported fatigue | Change from baseline to day 10 and day 21
  Patient self-reported fatigue using the scales PedsQL MFS (Child and adolescent versions) and FS-Adolescent and FS-Child, are exploratory endpoints.
Change in self-reported quality of life | Change from baseline to day 10 and day 21
  Patient self-reported quality of life using the scale PedsQL Acute Cancer Module (child and adolescent version) is another exploratory endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Schechter T, Tardif-Theriault C, Culos-Reed N, Lewis V, Orsey A, Diorio C, Tomlinson GA, Sung L. Yoga versus iPad active control for fatigue in paediatric cancer therapy: a randomised controlled trial. BMJ Support Palliat Care. 2025 Feb 26;15(2):204-212. doi: 10.1136/spcare-2023-004609. PMID 38160047